CLINICAL TRIAL: NCT07023822
Title: Women's Interventions for Sexual Health: WISH, Feasibility of a Factorial Design
Brief Title: WISH, Feasibility of a Factorial Design
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: UTK IRB-25-08813-XP
Record Dates: First submitted 2025-06-06; First posted 2025-06-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Vulvovaginal Signs and Symptoms; Sexual Desire Disorder; Body Image
Keywords: vulvovaginal atrophy; libido; hypnosis; progressive muscle relaxation
MeSH Terms: conditions — Breast Neoplasms | interventions — Histocompatibility Testing; Autogenic Training

STUDY DESIGN:
Intervention Model Description: This is a feasibility of a factorial design testing a multi-component intervention to improve vulvovaginal atrophy, sexual desire and body image. The investigators will also explore effect sizes of the chosen outcome measures to gather preliminary efficacy data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Hyaluronic acid (HLA) Vaginal Moisturizer + Hypnosis (Experimental): Participants will use an HLA vaginal moisturizer every 3 days, weeks 1-8.
  Participants will listen to hypnotic relaxation audio files at least 3x/week, weeks 3-8. There are 3 audio files in total, each about 20 min in length. The files are listened to in order. Each file is used for 2 weeks.
  Interventions: Device: Hyaluronic acid (HLA) Vaginal Moisturizer; Behavioral: Hypnotic Relaxation
- Hyaluronic acid (HLA) Vaginal Moisturizer + PMR (Experimental): Participants will use an HLA vaginal moisturizer every 3 days, weeks 1-8.
  Participants will listen to a progressive muscle relaxation (PMR) audio file at least 3x/week, weeks 3-8. There is only 1 PMR audio file. The same file will be used for 6 weeks.
  Interventions: Device: Hyaluronic acid (HLA) Vaginal Moisturizer; Behavioral: Progressive Muscle Relaxation (PMR)
- Hyaluronic acid (HLA) Vaginal Moisturizer Only (Experimental): Participants will use an HLA vaginal moisturizer every 3 days, weeks 1-8.
  Interventions: Device: Hyaluronic acid (HLA) Vaginal Moisturizer
- Polycarbophil Vaginal Moisturizer + Hypnosis (Experimental): Participants will use a polycarbophil vaginal moisturizer every 3 days, weeks 1-8.
  Participants will listen to hypnotic relaxation audio files at least 3x/week, weeks 3-8. There are 3 audio files in total, each about 20 min in length. The files are listened to in order. Each file is used for 2 weeks.
  Interventions: Device: Polycarbophil Vaginal Moisturizer; Behavioral: Hypnotic Relaxation
- Polycarbophil Vaginal Moisturizer + PMR (Experimental): Participants will use a polycarbophil vaginal moisturizer every 3 days, weeks 1-8.
  Participants will listen to a progressive muscle relaxation (PMR) audio file at least 3x/week, weeks 3-8. There is only 1 PMR audio file. The same file will be used for 6 weeks.
  Interventions: Device: Polycarbophil Vaginal Moisturizer; Behavioral: Progressive Muscle Relaxation (PMR)
- Polycarbophil Vaginal Moisturizer Only (Experimental): Participants will use a polycarbophil vaginal moisturizer every 3 days, weeks 1-8.
  Interventions: Device: Polycarbophil Vaginal Moisturizer

INTERVENTIONS:
Device: Hyaluronic acid (HLA) Vaginal Moisturizer — Use of vaginal moisturizer every 3 days for weeks 1-8.
  Arms: Hyaluronic acid (HLA) Vaginal Moisturizer + Hypnosis; Hyaluronic acid (HLA) Vaginal Moisturizer + PMR; Hyaluronic acid (HLA) Vaginal Moisturizer Only
Device: Polycarbophil Vaginal Moisturizer — Use of vaginal moisturizer every 3 days for weeks 1-8.
  Arms: Polycarbophil Vaginal Moisturizer + Hypnosis; Polycarbophil Vaginal Moisturizer + PMR; Polycarbophil Vaginal Moisturizer Only
Behavioral: Hypnotic Relaxation — Listen to hypnotic relaxation audio files at least 3x/week for weeks 3-8.
  Arms: Hyaluronic acid (HLA) Vaginal Moisturizer + Hypnosis; Polycarbophil Vaginal Moisturizer + Hypnosis
Behavioral: Progressive Muscle Relaxation (PMR) — Listen to PMR audio file at least 3x/week for weeks 3-8.
  Arms: Hyaluronic acid (HLA) Vaginal Moisturizer + PMR; Polycarbophil Vaginal Moisturizer + PMR

SUMMARY:
The primary aim of this study is to evaluate the feasibility of testing a multi-component intervention for sexual function using a factorial design.

DETAILED DESCRIPTION:
This proposal builds upon a multi-component pilot study (WISH), where women with a history of breast cancer participated in a two-component intervention to improve vulvovaginal atrophy with a vaginal moisturizer and sexual desire and body image with Hypnotic Relaxation (HR), a mind-body intervention that includes suggestions for relaxation, improved sexual desire, and body image delivered via audio file. This study seeks to further test WISH by expanding vulvovaginal atrophy interventions to include either a polycarbophil-based vaginal moisturizer (Replens™) or a hyaluronic acid-based moisturizer (HYALO GYN ®); and hypnosis relaxation (HR) or progressive muscle relaxation (PMR) interventions for sexual desire and body image. The primary outcome is the feasibility of a multi-component intervention for sexual function using a factorial design.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 female
2. Ability to read and write English
3. History of any stage of breast cancer
4. Completed primary treatment (chemotherapy, radiation and/or surgery) ≥3 months and ≤ 10 years prior to registration. Participants may use concurrent adjuvant endocrine therapy or HER2-targeted therapy while on study.
5. Able to engage in sexual activity including penetration or insertion into the vagina
6. Currently has a sexual partner.
7. Responds "yes" to "Do you currently experience vaginal or vulvar dryness and/or discomfort/pain with sexual activity?"
8. Responds "yes" to at least one of the following questions:

   * "Have you experienced negative changes in your body image since being diagnosed or treated for cancer?" or
   * "Have you experienced negative changes in your sexual desire since being diagnosed or treated for cancer?"

Exclusion Criteria:

1. Antidepressants are allowed if a person has been on them for 30 days prior to registration, and dose or treatment is not expected to change.
2. An active psychiatric disorder that is or causing you symptoms or distress, such as major depressive disorder, bipolar disorder, obsessive compulsive disorder, PTSD, schizophrenia or borderline personality disorder (Defined per medical history and/or patient self-report)
3. Currently enrolled in another study that addresses sexual health (enrollment in other clinical trials will be allowed).
4. Previous participant in WISH Study
5. Currently receiving active treatment
6. Use of oral, transdermal or vaginal estrogen
7. Allergy or intolerance to Replens, Hyalo Gyn or any of their components.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female at birth
Enrollment: 18 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Accrual Rate | Screening to consent, up to 30 days.
  The number of women who consented to participate in the study divided by the number who were eligible and educated about the study.
Retention Rate | Consent through study completion, an average of 8 weeks.
  The number of women who complete all 8 weeks of the study and complete the PROMIS SFS at baseline and at eight weeks divided by the number who are randomized and begin study treatment.
Adherence Rate, Moisturizer | Consent through study completion, an average of 8 weeks.
  The number of moisturizer uses completed by participants divided by the total number of possible moisturizer uses.
Adherence Rate, Relaxation Intervention | Consent through study completion, an average of 8 weeks.
  The number of times participant listened to assigned relaxation audio file (hypnosis or PMR) divided by the total number of possible listens.

OTHER OUTCOMES:
Exploratory Outcome, Female Sexual Function Index (FSFI) | Consent through study completion, an average of 8 weeks.
  The Female Sexual Function Index (FSFI) is a 19-item scale that measures the following domains of female sexual functioning, followed by subscale score ranges: desire (1.2-6), arousal (0-6), satisfaction (0.8-6), orgasm (0-6), lubrication (0-6) and pain (0-6). When the scores of these domains are added together, the sum represents an FSFI total score. The possible total score from 2-36 where higher scores indicate better sexual function.
Exploratory Outcome, PROMIS Sexual Function and Satisfaction (SFS) | Consent through study completion, an average of 8 weeks.
  The PROMIS scale is a 25 item measure that includes screener items. This study will include items asking about interest in sexual activity, lubrication, vaginal discomfort, vulvar discomfort, clitoral discomfort, orgasm and pleasure, and satisfaction. Raw scores must be converted to t-scores where the mean(standard deviation) = 50(10) in the referent population. Higher scores indicate more of the thing being described.
Exploratory Outcome, Breast Impact of Treatment Scale (BITS) | Consent through study completion, an average of 8 weeks.
  The BITS scale is a 13-item measure of body change stress in women with breast cancer. Possible scores range from 0-65 where higher scores indicate greater body change stress.
Exploratory Outcome, Sexual Distress Scale-Short Form (SDS-SF) | Consent through study completion, an average of 8 weeks.
  The SDS-SF is a 5-item scale that was developed based on the longer FSDS-R (Female Sexual Distress Scale, Revised). It is used to measure negative feelings like worry and frustration that people have about their sex lives and relationships. Possible scores range from 0-20. Higher scores indicate more of the thing being described.
Exploratory Outcome, Scale of Body Connection (SBC) | Consent through study completion, an average of 8 weeks.
  The SBC is a 20-item scale that measures two dimensions of body connection, body awareness (BSC-BA) measured with 12 items and bodily dissociation (SBC-BD) measured with 8 items. Possible scores for body awareness range from 0-48. Possible scores for the body dissociation range from 0-32. Higher scores indicate more of the thing being described.

CONTACTS AND LOCATIONS:
Overall Officials: Noel M Arrign, DNP, PhD, RN, Principal Investigator — College of Nursing, University of Tennessee
Locations (1):
- University of Tennessee, College of Nursing, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study and as such, data will be thoroughly interrogated. However, if a researcher feels there are unanswered questions or wishes to add to a larger dataset, the investigator would entertain all data-sharing requests for deidentified data as appropriate.